CLINICAL TRIAL: NCT01859403
Title: Nutrigenomics: Personalizing Weight Loss for Obese Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Amir Zarrinpar, MD, PhD, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VASDNUTRIMOVE13
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Obesity
Keywords: veteran; obesity; personalized genomics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Placebo Comparator): Usual care for veterans as part of the MOVE! program
  Interventions: Genetic: Usual Care
- Personalized Genomics (Active Comparator): Personalized genomics information from the FIT Test, Pathway Genomics
  Interventions: Genetic: Personalized Genomics

INTERVENTIONS:
Genetic: Personalized Genomics — A set of single nucleotide polymorphisms in genes important for obesity, eating behaviors and exercise
  Other Names: FIT test from Pathway Genomics, Inc.
  Arms: Personalized Genomics
Genetic: Usual Care — Patients receive the same dietary recommendation regardless of their genetic information
  Other Names: Standard dietary recommendations
  Arms: Usual Care

SUMMARY:
This study aims to determine if providing genomic information to veterans can help them lose weight compared to usual care.

DETAILED DESCRIPTION:
About 35% of veterans are obese. The MOVE! program is a nation-wide 8-week program of group classes nationally to help obese veterans lose weight. While the program is successful for some veterans, about 75% of veterans are unable to lose ≥5% of their weight 24 weeks after MOVE! New methods are needed to help obese veterans seeking weight loss. Using personalized genomic information dictating a specific diet, and information on exercise and eating behaviors, may be one means to help promote weight loss. Just a single nucleotide change or polymorphism (SNP) in a gene can increase a person's risk for obesity, or change their lipid profile in response to the consumption of different macronutrients such as of fats or carbohydrates. Over 54 genetic loci have been associated with obesity phenotypes and clinical studies are now reporting associations between SNPs and/or functional alterations of gene expression (epigenetics) and the ability to lose weight or not. We will implement a randomized clinical trial to test a set of genomic data called the FIT™ test (Pathway Genomics™) containing information on SNPs that affect obesity risk, confer specific diet recommendations, outline eating behaviors and suggest responses to various exercise regimens. The overall goal of this project is to evaluate if this supplemental genetic information with a genomically-derived diet built around packaged meals to improve adherence, in parallel with the MOVE! program at the VA in San Diego, will promote weight loss in more obese veterans than those receiving usual care and eating diets based around packaged meals. Our primary hypotheses are that more obese veterans in the MOVE! program will lose 5% of their weight if they receive personalized genomic information and a genomically-derived diet built around packaged meals when compared to veterans in the same program that receive usual care during MOVE! and packaged meals after 8 or 24 weeks. We also hypothesize that more veterans in the genomic group that lose 5% weight loss at 8 weeks will maintain this weight loss after 24 weeks compared to veterans in the usual care group.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans able to receive care at the VASDHS and planning to start the MOVE! program.
2. Veterans able to understand and consent to the study.
3. BMI equal to or greater than 30 kg/m2.

Exclusion Criteria:

1. Veterans unable to receive care at the VASDHS.
2. Veterans unable to understand the consent process at the discretion of the PI.
3. Active substance abuse or substance dependence disorder
4. Cognitive disorder, psychiatric hospitalization in past 6-months, or presence of suicidal ideation identified on self-report instruments
5. Bradycardia, rapid heart rate or other arrhythmia or active ischemia by EKG.
6. Uncontrolled thyroid disease as measured by a TSH above or below the normal range.
7. Body mass index < 30 kg/m2.
8. Chronic kidney disease stage III or higher by National Kidney Foundation criteria (GFR = 30-59 ml/min).
9. New York Heart Association's functional classification of congestive heart failure above Class I (not limited with normal physical activity by symptoms; Class II occurs when ordinary physical activity results in fatigue, dyspnea, or other symptoms).
10. Sodium or potassium outside the normal range.
11. Edema requiring the use of daily diuresis with furosemide, bumex or other diuretic (does not include hydrochlorthiazide).
12. The use of high dose oral corticosteroids (above replacement doses).
13. Veterans deficient in 25-OH vitamin D (<20 units/dl).
14. Veterans with fasting LDL > 190 mg/dl.
15. Veterans with fasting triglyceride levels > 1000 mg/dl.
16. Excessive caffeine use (>6 caffeinated beverages/days).
17. Prior gastrointestinal surgery with the exception of distal appendectomy.
18. Acute infections or current use of antibiotic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

REFERENCES:
- [Derived] Frankwich KA, Egnatios J, Kenyon ML, Rutledge TR, Liao PS, Gupta S, Herbst KL, Zarrinpar A. Differences in Weight Loss Between Persons on Standard Balanced vs Nutrigenetic Diets in a Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2015 Sep;13(9):1625-1632.e1. doi: 10.1016/j.cgh.2015.02.044. Epub 2015 Mar 10. PMID 25769412

RESULTS

PARTICIPANT FLOW:
Period: Primary Endpoint Measure
Arm/Group | Usual Care | Personalized Genomics
Started | 21 | 30
Completed | 20 | 26
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 0 | 1
Period: Secondary Endpoint Measure
Arm/Group | Usual Care | Personalized Genomics
Started | 20 | 26
Completed | 14 | 18
Not Completed | 6 | 8
Not completed — Withdrawal by Subject | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Personalized Genomics | Total
Number analyzed (Participants) | 20 | 26 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (12.3) | 48.4 (13.1) | 51.1 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 17 | 16 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 13 | 12 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 20 | 26 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Weight Loss of 5% or More at 8 Weeks
Description: Our primary hypotheses are that more obese veterans in the MOVE! program will lose greater or equal to 5% of their weight if they receive personalized genomic information and a genomically-derived diet built around packaged meals when compared to veterans in the same program that receive usual care during MOVE! and packaged meals after 8 weeks.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Personalized Genomics
Number analyzed (Participants) | 20 | 26
Participants | 7 | 7

2. Secondary Outcome: Number of Participants With Weight Loss of 5% or More at 24 Weeks
Description: We hypothesize that more veterans in the genomic group that lose greater or equal to 5% weight loss at 8 weeks will maintain this weight loss after 24 weeks compared to veterans in the usual care group.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Personalized Genomics
Number analyzed (Participants) | 14 | 18
Participants | 5 | 7

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Usual Care | Personalized Genomics
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/26
Other Adverse Events (participants affected / at risk) | 0/20 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No